CLINICAL TRIAL: NCT04365439
Title: Convalescent Plasma for the Treatment of Moderate-severe COVID-19: A Proof-of-principle Study
Brief Title: Convalescent Plasma for COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Enos Bernasconi (Other)
Responsible Party: Sponsor-Investigator, Enos Bernasconi, Prof Dr med, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-00895
Record Dates: First submitted 2020-04-18; First posted 2020-04-28 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Blood Plasma Therapy; COVID

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Convalescent plasma (Experimental): Convalescent plasma from patients after COVID-19
  Interventions: Biological: Blood plasma

INTERVENTIONS:
Biological: Blood plasma — Convalescent plasma after COVID-19

SUMMARY:
The purpose of this proof of concept study is to provide COVID-19 convalescent plasma to patients with moderate to severe COVID-19 and assess:

* the titer of anti-COVID-19 antibodies in the donors and in the patients before and after treatment;
* the in-depth analysis of immunological parameters in the donors and in recipient before and after treatment;
* the impact of plasma transfusion on the reduction of viral load and inflammation
* safety and tolerability
* clinical efficacy

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized adult patients 18 - 75 y.o. with confirmed COVID-19 infection by nasopharyngeal swab;
* radiologically confirmed pneumonia;
* SpO2 > 92o/o and < 96% (room air);
* ongoing thromboembolic prophylaxis.

Exclusion Criteria:

* Participation to another COVID-19 trial;
* severe COVID-19 disease (SpO2 < 93o/o in room air);
* severe allergic transfusion reactions or anaphylaxis in the patient history;
* documented lgA deficiency;
* unstable heart disease with signs of circulatory overload;
* malignancies or other concomitant diseases with poor short-term prognosis;
* pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Titers of anti-SARS-CoV-2 antibodies in the plasma derived from convalescent donors | At plasma donation
Change in titers of anti-SARS-CoV-2 antibodies in patients' plasma | Change from baseline at day 21
Change in inflammatory cytokines concentration (e.g. IL-6, HMGB1) | Change from baseline at day 7
Viral load decay in the recipient after plasma transfusion with semiquantitative assessment of nasopharyngeal swabs | Change from day of diagnosis at day 1
  Semiquantitative measure of viral load by rtPCR for SARS-CoV-2 by nasopharyngeal swabs, at diagnosis and on day 1,3,7

SECONDARY OUTCOMES:
Number of patients with improvement in the 7-points Ordinal Scale | At day 7
  7-point ordinal scale measure on day 0 (Baseline), day 1, 3 and 7 after plasma transfusion
Proportion of patients with adverse events, severity of adverse events | At day 21
  AE will be assessed by the DAIDS scale on day 1, 3, 7 and 21. Relatedness with plasma transfusion will also be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Fontana, M.D., Principal Investigator — Servizio Trasfusionale, Lugano
Locations (1):
- Ospedale Regionale Locarno, Locarno, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shen C, Wang Z, Zhao F, Yang Y, Li J, Yuan J, Wang F, Li D, Yang M, Xing L, Wei J, Xiao H, Yang Y, Qu J, Qing L, Chen L, Xu Z, Peng L, Li Y, Zheng H, Chen F, Huang K, Jiang Y, Liu D, Zhang Z, Liu Y, Liu L. Treatment of 5 Critically Ill Patients With COVID-19 With Convalescent Plasma. JAMA. 2020 Apr 28;323(16):1582-1589. doi: 10.1001/jama.2020.4783. PMID 32219428